CLINICAL TRIAL: NCT00795899
Title: Preoperative Therapy With Epirubicin/Cyclophosphamide Followed by Paclitaxel/Trastuzumab and Postoperative Therapy With Trastuzumab in Patients With HER-2 Over Expressed Breast Cancer
Brief Title: Taxol Epirubicin Cyclophosphamide Herceptin Neoadjuvant (TECHNO)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GBG Forschungs GmbH (Other)
Collaborators: AGO Study Group (Other)
Responsible Party: Udo Pfeil, GBG Forschungs GmbH
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TECHNO
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2011-08

CONDITIONS: Breast Cancer
Keywords: Safety and efficacy of experimental treatment
MeSH Terms: conditions — Breast Neoplasms | interventions — Epirubicin; Cyclophosphamide; Paclitaxel; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Epirubicin/Cyclophosphamide in combination with Paclitaxel/Trastuzumab, followed by postoperative Trastuzumab in patients with HER-2 overexpression
  Interventions: Drug: Epirubicin / Cyclophosphamide in combination with Paclitaxel/Trastuzumab, followed by postoperative Trastuzumab

INTERVENTIONS:
Drug: Epirubicin / Cyclophosphamide in combination with Paclitaxel/Trastuzumab, followed by postoperative Trastuzumab — Cycles 1-4 Epirubicin: 90 mg/m2, i.v. day 1 Cyclophosphamide: 600 mg/m2, i.v. day 1 Every 22d
  Cycles 5-8 Paclitaxel: 175 mg/m2, i.v., 3h-infusion day 1 Trastuzumab: 8 mg/kg i.v. at day 0 of the 5th cycle and thereafter each 6 mg/kg i.v. day 1 in the cycles 6-8 Every 22d

SUMMARY:
The present clinical trial will investigate the safety and efficacy of a sequential preoperative therapy with Epirubicin/Cyclophosphamide in combination with Paclitaxel/Trastuzumab, followed by postoperative Trastuzumab in patients with HER-2 overexpression primary breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Primary carcinoma of the breast, confirmed histologically by core biopsy (at least 3 core biopsy samples)
2. Tumor lesion of the breast with a palpable or a imagistic size ≥ 2 cm or inflammatory breast cancer
3. Known HER-2 status detected on core biopsy. HER-2 over expression is defined as DAKO HercepTest (3+) or DAKO HercepTest (2+) and FISH (+) (fluorescence-in-situ-hybridisation).
4. No distant metastatic disease, confirmed by chest x-ray, abdominal sonography and bone scan.
5. Female patients
6. Age ≥ 18 and ≤ 65 years
7. ECOG < 2/WHO 0-1
8. Laboratory requirements GOT and Bilirubin < 1.5x UNL Leukocytes >= 3 G/l Neutrophile > 1 G/l Thrombocytes > 100 G/l Creatinine (Serum) < 2.0 mg/dl.
9. Normal cardiac function, confirmed by cardiologist
10. No active hepatitis
11. Written informed consent for all study procedures
12. Patients must be available and compliant for treatment and follow-up

Exclusion Criteria:

1. Multicentricity in various quadrants (contact the study office)
2. CNS-metastases
3. Secondary malignancy, excluding basalioma of the skin or carcinoma in situ of the cervix that has received curative therapy
4. Patients with relevant hemodynamic cardial diseases
5. Patients with a left ventricular ejection fraction (LVEF) under the normal limit of the institution, confirmed by echocardiography or MUGA-Scan.
6. Uncontrolled, severe comorbidities
7. Patients with severe respiratory diseases and severe dyspnea and / or which need supportive oxygen
8. Previous anti-HER2-therapy
9. Patients receiving immunosuppressant therapy
10. Known allergy to medication containing cremophor
11. Hb <10 g/dL, Neutrophile <1.5 x109/L, Thrombocytes <100 x109/L.
12. Total-Serum-Bilirubin >1.5 x ULN (upper limit of normal) (except in patients with confirmed and documented Gilbert-Lereboullet-syndrome), ALT or AST >2.5 x ULN (>5 x ULN by liver metastases), Alkaline Phosphatase >2.5 x ULN (>4 x ULN by liver or bone metastases), Serumcreatinine > 2 x ULN
13. Pregnancy, nursing (a negative pregnancy test must be documented, and safe anticontraceptive measures during pre- and postoperative treatment must be implemented)
14. Lack of signed informed consent after informing the patient
15. Lack of willingness to keep and disclose personal medical data as part of the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2002-01; Primary Completion 2005-12 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To estimate the rate of cardiac (serious) events NYHA III/IV-and pathological complete remission after study therapy. | 36 months

SECONDARY OUTCOMES:
To assess: the rate of breast conserving surgery, the clinical response rates, the histopathological lymph node status after preoperative therapy, the disease-free and overall survival. | 36 months
To evaluate the quality of life. | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Untch, MD, Prof., Principal Investigator — AGO Study Group
Locations (1):
- Ludwig Maximillian University Munich, Department of Gynecology and Obstetrics, Munich, Bavaria, Germany

REFERENCES:
- [Derived] von Minckwitz G, Untch M, Blohmer JU, Costa SD, Eidtmann H, Fasching PA, Gerber B, Eiermann W, Hilfrich J, Huober J, Jackisch C, Kaufmann M, Konecny GE, Denkert C, Nekljudova V, Mehta K, Loibl S. Definition and impact of pathologic complete response on prognosis after neoadjuvant chemotherapy in various intrinsic breast cancer subtypes. J Clin Oncol. 2012 May 20;30(15):1796-804. doi: 10.1200/JCO.2011.38.8595. Epub 2012 Apr 16. PMID 22508812